CLINICAL TRIAL: NCT02679339
Title: A Phase Ib Pilot Multiple Dose, Randomized-Withdrawal, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Pharmacokinetics of Topically Applied 40% Lidocaine Gel Compared With Placebo in Subjects With Acute Herpes Zoster Pain
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Topically Applied 40% Lidocaine Gel Compared With Placebo in Subjects With Acute Herpes Zoster (Shingles) Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Limited patient enrollment
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-HZ-011
Record Dates: First submitted 2015-02-09; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Acute-onset Herpes Zoster Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CNTX-2022 (lidocaine gel, 40%) (Experimental): Application of 1mL CTNX-2022 (40% Anhydrous Lidocaine Gel) topically applied to 300cm squared outlined area once daily (in the morning) for 8 days at the study site.
  Interventions: Drug: CNTX-2022 (lidocaine gel, 40%)
- Placebo (Placebo Comparator): Application of 1mL placebo topically applied to 300cm squared outlined area once daily (in the morning) for 8 days at the study site.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTX-2022 (lidocaine gel, 40%)
  Arms: CNTX-2022 (lidocaine gel, 40%)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study 2022-HZ-011 will utilize a randomized withdrawal (RW), double-blind, placebo controlled design in which the PK and safety of CNTX 2022 (40% anhydrous lidocaine gel) will be evaluated in subjects with acute-onset herpes zoster pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female ≥ 18 years of age and ≤ 85 years of age.
2. Subject has brush-evoked allodynic pain intensity score ≥ 4 using the NPRS as determined by pain assessment during the physical examination at screening.

   a. Onset must have occurred ≤ 20 days prior to randomization
3. Subject has an average daily pain intensity score of ≥ 4 using the NPRS as determined by pain assessment during the physical examination at screening.
4. Subject must have a diagnosis of herpes zoster (shingles).
5. Subject has rash limited to trunk and limbs, with a total surface area of up to 300 cm2.

Exclusion Criteria:

1. Subject has an active herpes zoster lesion on the face, head, neck, genital or rectal areas.
2. Subject has rash limited to trunk and limbs, with a total surface area greater than 300 cm2.
3. Subject has a known history of allergic reaction, hypersensitivity, or clinically significant intolerance to lidocaine, ingredients of the study drug, or local anesthetics of the amide type.
4. Subject has target skin area (allodynic area and surrounding skin) that is not intact, is inflamed, or in the opinion of the Principal Investigator, consistent with rash due to acute herpes zoster.
5. Subject has any other form of pain that was not discernible from herpes zoster (shingles) allodynia.
6. Subject is taking Class I antiarrhythmic drugs (e.g., tocainide, mexiletine), or medications that could interact with the study drug or interfere with its evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of topically applied 40% lidocaine gel measuring incidence, intensity, relationship, and seriousness of treatment-emergent AEs | 28 days
To evaluate the pharmacokinetics of topically applied 40% lidocaine gel measuring Tmax | 28 days

SECONDARY OUTCOMES:
To assess the effect of 40% lidocaine gel on 0-10 numeric pain rating scale (NPRS) scores related to acute herpes zoster | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Araco, MD, Principal Investigator — Nucleus Network Melbourne, Australia
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia